CLINICAL TRIAL: NCT06875193
Title: Key Finding of DM Treatment with Combination, a MuLticenter, Randomized, Parallel, Gathering Information of Phase 4 Trial to Evaluate the Efficacy and Safety of Dapagliflozin or Pioglitazone Add-on to Metformin and DPP-4 Inhibitor in Patients with Type 2 Diabetes
Brief Title: DM Treatment to Evaluate the Efficacy and Safety of Dapagliflozin or Pioglitazone in Patients with Type 2 Diabetes
Acronym: KLIMT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DW6012-IV-2
Record Dates: First submitted 2025-02-24; First posted 2025-03-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Type2diabetes
Keywords: Dapagliflozin; Pioglitazone; DPP-4 inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dasidiem 10/100mg (Experimental): Dapagliflozin 10mg +sitagliptin 100mg combination drug
  Interventions: Drug: DW6012(Dasidiem tab. 10/100mg)
- sitdiem 100mg, Piotazone15mg (Active Comparator): sitagliptin 100mg, Pioglitazone 15mg
  Interventions: Drug: DW6012(Dasidiem tab. 10/100mg)

INTERVENTIONS:
Drug: DW6012(Dasidiem tab. 10/100mg) — Once a day, Oral administration
  Other Names: Piotazone tab.; Sitdiem tab. 100mg

SUMMARY:
Key finding of DM Treatment with combination, A MuLticenter, Randomized, Parallel, Gathering Information of phase 4 Trial to Evaluate the Efficacy and Safety of Dapagliflozin or Pioglitazone add-on to Metformin and DPP-4 inhibitor in Patients with Type 2 Diabetes Who Have Inadequate Glycaemic Control on a Background Combination of Metformin and DPP-4 inhibitor(KLIMT Study)

DETAILED DESCRIPTION:
This is a Phase 4, multicenter, randomized, open-label, parallel clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes who are 19 years of age or older at the date of written consent
* Subjects who Receiving a stable dose of metformin and a DPP-4 inhibitor for at least the last 8 weeks at the time of screening
* HbA1c ≤ 7.0% ≤ HbA1c < 10% at time of screening
* BMI ≤ 18.5 kg/m2 ≤ 40 kg/m2 at time of screening
* Subjects fully explained and understood the purpose and methods of this study and voluntarily gave written informed consent

Exclusion Criteria:

* Patients with type 1 diabetes
* Have a BMI > 40 kg/m2
* Subjects who have moderate (Stage 3b) or severe kidney disease or an estimated glomerular filtration rate (eGFR, using the CKD-EPI formula) < 45 mL/min/1.73 m2
* Patients with end stage renal disease or patients on dialysis
* Patients with uncontrolled heart failure (NYHA class III - IV)
* Patients with history of uncontrolled arrhythmia, myocardial infarction, unstable angina, coronary artery bypass graft surgery, cerebrovascular disease within 24 weeks prior to the screening visit
* Patients with acute or chronic metabolic acidosis, including lactic acidosis, diabetic ketoacidosis (DKA) with or without coma, and patients with a history of ketoacidosis
* Patients with diabetic coma or precoma
* Patients with a history of severe hypoglycemia while taking metformin and DPP-4 inhibitors.
* Patients with hematuria
* Patients who receiving treatment for thyroid dysfunction at the time of screening
* Malnourished, starving, or debilitated subjects
* Patients with pituitary insufficiency or adrenal insufficiency
* Patients with clinically significant hepatic disease with AST or ALT greater than 3 times the upper limit of normal
* Patients with severe infectious diseases, perioperative, or clinically significant trauma
* Have a history of substance abuse
* Patients receiving insulin or sulfonylurea, thiazolidinedione, SGLT2 inhibitor, GLP-1 receptor agonist within 8 weeks prior to the screening visit
* Patients who have received more than 2 consecutive weeks of corticosteroids within 8 weeks at the time of screening or who require treatment requiring repeated use of corticosteroids
* Patients with a history of malignancy within the last 5 years
* Participation in any other clinical trial within 12 weeks of screening in which an investigational drug or investigational medical device was administered or applied
* Pregnant and breastfeeding women
* Hypersensitivity to any of the drugs and components, including metformin, DPP-4 inhibitors, dapagliflozin, TZDs, sulfonylurea class of drugs, or any of the ingredients
* Patients with genetic problems such as galactose intolerance, Lapp lactose deficiency, or glucose-galactose mal-absorption.
* Any other person deemed by the investigator to be unsuitable for participation in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Variance in HbA1c from baseline to 24 weeks on study drug | 24 weeks
  Change in HbA1c

SECONDARY OUTCOMES:
Variance in HbA1c from baseline to 12 weeks on study drug | 12 weeks
  Change in HbA1c
Variance in FPG from baseline to 12, 24 weeks on study drug | 12, 24 weeks
  Change in Fasting Plasma Glucose(FPG)
Variance in TC(mg/dL), TG(mg/dL), HDL(mg/dL), LDL(mg/dL) from baseline to 12, 24 weeks on study drug | 12, 24 weeks
  Change in TC, TG, HDL, LDL
Variance in FLI(Fatty Liver Index), AST, ALT, r-GTP, ALP, HSI(Hepatic steatosis index), Total bilirubin, Albumin, Protein from baseline to 12 and 24 weeks after study drug administration | 12, 24 weeks
  FLI(Fatty Liver Index)= 1/(1+exp(-x))×100
  HSI(Hepatic steatosis index) = 8×ALT/AST+BMI(+2, if type 2 diabetes yes, +2 if female)
Variance in Kidney value from baseline to 12, 24 weeks on study drug | 12, 24 weeks
  Kidney value: eGFR(CKD-EPI fomulation) ACR(Albumin to Creatine ratio), Creatinine
Variance in body weight from baseline to 12, 24 weeks on study drug | 12, 24 weeks
Percentage of patients achieving HbA1c of 7.0% or 6.5% or less at 12 and 24 weeks post study drug administration compared to baseline | 12, 24 weeks
  Percentage of patients achieving HbA1c of 7.0% or 6.5% or less
Variance in Insulin from baseline to 12, 24 weeks on study drug | 12, 24 weeks
Percentage of subjects prescribed an rescue drug during this study | during 24weeks(study duration/per subject)
  rescue drug
Variance in waist measurement from baseline to 12, 24 weeks on study drug | 12, 24 weeks
Variance in BMI from baseline to 12, 24 weeks on study drug | 12, 24 weeks
Variance in blood pressure from baseline to 12, 24 weeks on study drug | 12, 24 weeks
Variance in HOMA-IR, HOMA-β(Glucose in Molar Units mmol/L) from baseline to 12, 24 weeks on study drug | 12, 24 weeks
Variance in c-peptide from baseline to 12, 24 weeks on study drug | 12, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No